CLINICAL TRIAL: NCT00535990
Title: Minimally Invasive Surgery (MIS) Database Looking at Patterns of Care, Outcomes, and Prognostic Analysis for the Purpose of Research
Brief Title: Minimally Invasive Surgery (MIS) Database for the Purpose of Research
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Santiago Horgan, Professor of Surgery, University of California, San Diego
Other Study IDs: 070449; Internally funded
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Morbid Obesity; Hernia; Colorectal Cancer; Laparoscopy
Keywords: Cholecystectomy; Appendectomy; Esophageal; Surgical; Procedures; Surgery; Gastric; bypass
MeSH Terms: conditions — Obesity, Morbid; Hernia; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Minimally Invasive Surgery Team (MIST) are establishing a separate research database to find out more about patient's undergoing minimally invasive surgery (laparoscopic , open and robot assisted) procedures at UCSD. The hope is that collection of this information will give physicians a better knowledge and understanding of the benefits of minimally invasive surgery and possibly assist physicians to better manage future patients.

DETAILED DESCRIPTION:
Minimally invasive surgery has become the gold standard in surgical treatment for many indications, such as treatment of gallstones and acute appendicitis. For many other indications, the potential for minimally invasive approaches exist, but the data does not yet exist to establish it as the gold standard. In addition, there are certain patient factors such as age or weight that may influence the success of a minimally invasive procedure.

While there are numerous articles in the literature reporting outcomes for minimally invasive therapies, these series are often notable for small patient populations and varying definitions of treatment success from study to study. Due to the lack of uniformity in reporting patient outcomes, an opportunity exists to establish a standardized database of a large number of patients undergoing these procedures.

A standardized database will facilitate conducting prospective research of the risk factors and benefits of minimally invasive surgery. This analysis will not only enhance the care provided to these patients, it will reduce the use of ineffective therapy, thus promoting improved efficiency while increasing the quality of care provided within the UCSD system.

This is our initial application. Several other departments at UCSD have developed similar databases. There are numerous examples of prospective databases used for similar purposes in the literature. Smithers, et al, used a prospective database of 446 patients undergoing esophagectomy to compare open to laparoscopic outcomes. Nesset, et al, maintained a database of bariatric surgery patients for two decades and was able to draw conclusions from a data set of 1584 patients. Even at smaller numbers, a prospective database is useful. Andrew, et al, described the improvement in outcomes over the learning curve in the first 201 patients undergoing laparoscopic roux-en-Y gastric bypass using such a database. Though labor intensive, Clemmesen, et al, found maintaining a database allowed them to improve care for their patients.

ELIGIBILITY:
Inclusion Criteria:

Gastric Banding Group:

* For gastric banding subjects to qualify for study inclusion, subjects have to have a BMI ranging from 33-40. Currently a BMI of 33 is our lower level of acceptable for bypass.

Control Group:

* All adult subjects 18 years or greater being seen in the minimally invasive surgery clinic for elective laparoscopic surgery will also be screened.

Exclusion Criteria:

* Subjects with a BMI>40 will be excluded because their fat cells are very large and therefore fragile and unsuitable for research use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All male and female patients undergoing surgery at this center for either obesity surgery or for miimally invasive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Horgan, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgical Intervention: All patients in the minimally invasive surgery database are patients who have undergone surgical intervention by the Minimally Invasive Surgery faculty. Patients can be further stratified based on the type of procedure that they received. Since this study is primarily creation of a comprehensive database, patient's are not intentionally placed in a certain study arm aside from their procedure type.
Period: Overall Study
Arm/Group | Surgical Intervention
Started | 250
Completed | 250
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Surgical Intervention
Number analyzed (Participants) | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 175
  >=65 years | 75
Age, Continuous [Mean (Full Range); unit: years] | 57 [25 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 138

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Outcomes
Description: Post-operative outcomes including:
  30 day morbidity 30 day mortality 30 day readmission Surgical site infection Surgical site occurrences Surgical Reintervention Specific Surgical outcomes (staple line leak, etc)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Surgical Intervention
Number analyzed (Participants) | 250
participants
  30 day morbidity | 27
  30 day mortality | 0
  30 day readmission | 6
  surgical site infection | 4

ADVERSE EVENTS:
Arm/Group | Surgical Intervention
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes